CLINICAL TRIAL: NCT05405595
Title: A Phase 1b/2, Open-Label, Dose Escalation and Expansion Study of ADG126 in Combination With Pembrolizumab (Anti PD-1 Antibody) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: ADG126 in Combination With Pembrolizumab in Patients With Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adagene Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG126-P001; KEYNOTE-C98, MK-3475-C98 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-05-16; First posted 2022-06-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced/Metastatic Solid Tumors
Keywords: ADG126-P001
MeSH Terms: interventions — pembrolizumab; Standard of Care; Trifluridine; trifluridine tipiracil drug combination; Bevacizumab; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ADG126 in combination with Pembrolizumab (Trade name KEYTRUDA®) (Experimental): An IV infusion of ADG126 over 60-90 minutes will be administered 30-60 minutes after administration of pembrolizumab (KEYTRUDA®) infusion. A treatment cycle will consist of 21 days. ADG126 and Pembrolizumab (KEYTRUDA®) combination treatment both will be dosed until progressive disease (PD), intolerable toxicities, withdrawals of consent, or up to 35 cycles.
  Interventions: Drug: ADG126; Drug: Pembrolizumab (KEYTRUDA®)
- ADG126 and pembrolizumab (KEYTRUDA®) in combination with Trifluridine/Tipiracil-Bevacizumab (Experimental): To evaluate the preliminary antitumor efficacy of ADG126 and Pembrolizumab (KEYTRUDA®) in combination with SOC (Trifluridine/Tipiracil-Bevacizumab) while assessing safety and tolerability. Standard of care treatment will be administered according to the specifications outlined in the Investigational Brochure. Will be dosed until progressive disease (PD), intolerable toxicities, withdrawals of consent, or up to 35 cycles.
  Interventions: Drug: ADG126; Drug: Pembrolizumab (KEYTRUDA®); Drug: Standard of Care (Trifluridine/Tipiracil-Bevacizumab)
- ADG126 and pembrolizumab (KEYTRUDA®) in combination with fruquintinib (Experimental): To evaluate the preliminary antitumor efficacy of ADG126 and Pembrolizumab (KEYTRUDA®) in combination with SOC (Fruquintinib) while assessing safety and tolerability. The dose strength for treatment will be based on the IB and protocol. Fruquintinib (Fruzaqla) is orally given once daily for the first 21 days of each 28-day cycle. Each treatment cycle consists of 14 days. Will be dosed until progressive disease (PD), intolerable toxicities, withdrawals of consent, or up to 35 cycles.
  Interventions: Drug: ADG126; Drug: Pembrolizumab (KEYTRUDA®); Drug: Standard of care (Fruquintinib)
- Dose Optimization (Experimental): The randomized phase 2 Dose Optimization arm is intended to test two dosing regimens of ADG126 in combination with pembrolizumab (KEYTRUDA®), which allows the selection of an optimal regimen. The study treatments may continue for up to 35 treatments for pembrolizumab (KEYTRUDA®) if given every 21 days and 18 treatments for pembrolizumab (KEYTRUDA®) if given every 42 days until PD, intolerable toxicities or withdrawal of consent.
  Interventions: Drug: ADG126; Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: ADG126 — ADG126 is an anti-CTLA-4 fully human monoclonal antibody that specifically binds to human CTLA-4.
Drug: Pembrolizumab (KEYTRUDA®) — Pembrolizumab (KEYTRUDA®) is a PD-1 receptor-blocking antibody (a humanized IgG4 monoclonal antibody).
  Other Names: KEYTRUDA®
Drug: Standard of Care (Trifluridine/Tipiracil-Bevacizumab) — The standard of care therapies will include Trifluridine/Tipiracil-Bevacizumab, approved for treating metastatic colorectal cancer (CRC)and various solid tumors.
  Other Names: Lonsurf and Avastin
  Arms: ADG126 and pembrolizumab (KEYTRUDA®) in combination with Trifluridine/Tipiracil-Bevacizumab
Drug: Standard of care (Fruquintinib) — The standard of care therapy, Fruquintinib, is approved for treating metastatic colorectal cancer (CRC) and various solid tumors.
  Other Names: Fruzaqla
  Arms: ADG126 and pembrolizumab (KEYTRUDA®) in combination with fruquintinib

SUMMARY:
This is a Phase 1b/2, open-label, dose escalation, dose expansion and dose optimization study to evaluate the safety, tolerability, PK, and immunogenicity of ADG126-pembrolizumab combination regimens in patients with advanced/metastatic solid tumors.

The study drug ADG126 is an anti-CTLA-4 fully human monoclonal antibody that specifically binds to human CTLA-4. Pembrolizumab is a PD-1 receptor-blocking antibody (a humanized IgG4 monoclonal antibody).

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, multicenter, dose escalation, dose expansion and dose optimization study to evaluate the safety, tolerability, PK, and preliminary efficacy of ADG126-Pembrolizumab or ADG126-Pembrolizumab in combination with trifluridine/tipiracil-bevacizumab or fruquintinib in patients with advanced/metastatic solid tumors, with a focus on MSS CRC.

In Phase 2, the study will use a randomized design to evaluate the dose optimization regimen in patients with MSS CRC for ADG126- Pembrolizumab doublet only.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
3. Wash out period from previous antitumor therapies
4. At least 1 measurable lesion at baseline according to the definition of RECIST v1.1.
5. Adequate organ function.
6. An archival tumor biopsy is required and should be taken within 2 years of enrollment. If not available, a fresh tumor biopsy is acceptable.
7. For Dose Escalation Phase Only: Patients with histologically or cytologically confirmed, locally advanced or metastatic solid tumors, who have progressed after all standard therapies, or for whom no further standard therapy exists.
8. Dose Expansion Phase Only: Tumor tissues (archived tissue) before treatment are required for all patients.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Childbearing potential who does not agree to the use of contraception during the treatment period.
3. Treatment with any investigational drug within washout period.
4. Prior treatment with a PD-1, PD-L1 targeting agent or a next-generation anti-CTLA-4 therapy with enhanced ADCC function.
5. History of significant irAEs or irAE.
6. Central nervous system (CNS) disease involvement.
7. History or risk of autoimmune disease.
8. Patients requiring systemic treatment with corticosteroids or other immunosuppressive medications (>10 mg/day prednisone or equivalent).
9. Any uncontrolled active infections requiring systemic antimicrobial treatment (viral, bacterial, or other), or uncontrolled or poorly controlled, asthma, chronic obstructive pulmonary disease (COPD).
10. Major surgery within 4 weeks prior to the first dose of the study drug.
11. Has had an allogeneic tissue/solid organ transplant.
12. Has received a COVID-19 vaccine within 7 days prior to the first dose of study treatment. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Administration of killed vaccines are allowed.
13. A positive COVID-19 test within 14 days of Cycle 1 Day 1.
14. History of Hypersensitivity or known to be allergic to protein drugs or recombinant protein.
15. Active hemoptysis or central airway invasion by metastatic tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and RP2D for ADG126 in combination with pembrolizumab. | 9 months
  To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) for ADG126+ pembrolizumab in dose escalation levels
the safety and tolerability of ADG126 at escalating dose level in combination with pembrolizumab in adults with advanced metastatic solid tumors | 9 months
  Incidence rate of AEs as assessed by CTCAE v5.0
Access the preliminary antitumor activity of ADG126-pembrolizumab combination regimens | 9 months
  Number of Participants with preliminary antitumor activity
Maximum tolerated dose (MTD) and/or RP2D for ADG126 with Trifluridine/Tipiracil-Bevacizumab | 6 months
  To assess the safety and tolerability of ADG126 + pembrolizumab in combination with the following SOC therapies (Trifluridine/tipiracil-bevacizumab) in MSS CRC
  To determine the MTD and/or RP2D for ADG126 + pembrolizumab in combination with the following SOC therapies in MSS CRC:
Access the preliminary antitumor activity of ADG126 with Pembrolizumab in combination standard of care | 6 months
  To assess the preliminary antitumor activity of ADG126 + pembrolizumab in combination with the following SOC therapies in MSS CRC (Trifluridine/tipiracil-bevacizumab)
  SOC (Fruquintinib)
Access and characterize the optimal dose based on safety and efficacy parameters | 9 months
  To characterize the optimal dose based on safety and efficacy parameters

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile/parameters | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  Area under the time concentration curve (AUC) from time zero to infinity (AUC0-inf)
Maximum (peak) plasma concentration (Cmax) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  Maximum (peak) plasma concentration (Cmax)
Time to maximum (peak) concentration (Tmax) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  Time to maximum (peak) concentration (Tmax)
Trough concentration (Ctrough) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  Trough concentration (Ctrough)
Incidence of ADAs | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  this will be summarized for all patients who received at least 1 administration of ADG126. efficacy and safety will be evaluated.
To assess the disease control rate (DCR) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  this will be calculated as the proportion/percentage of patients with best overall response of CR,PR,SD or progressive disease will be calculated.
To assess the progression free survival (PFS) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  PFS will be censored at the time of the last evaluable tumor assessment (RECISTv1.1 and iRECIST)
To assess the overall survival (OS) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  This will be used to estimate median survival times where applicable.
To assess the efficacy outcomes in the defined patient population | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
  The dose optimization arm will be used to access the efficacy outcome derived in the defined patient population

CONTACTS AND LOCATIONS:
Overall Officials: Jiping Zha, MD, PhD, Study Director — Adagene Inc
Locations (21):
- United States (7):
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County, Irvine, California
  - Florida cancer specialist/Sarah Cannon Research Institute, Sarasota, Florida
  - The Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- China (4):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - SunYat-Sen University Cancer Center, Guangzhou, Guangdong
  - Hong Kong Humanity & Health Clinical Trial Center, Hong Kong, Hong Kong
  - Prince of Wales Hospital, Hong Kong, Hong Kong
- South Korea (10):
  - Dong -A University Hospital, Seogu, Busan Gwangyeogsi
  - CHA Bundang Medical Center, CHA university, Seongnam, Gyeonggido
  - The Catholic University of Korea Street. Vincent Hospital, Suwon, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - KangBuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No